CLINICAL TRIAL: NCT05174871
Title: Time-Restricted Feeding in Children and Adolescents With Obesity
Acronym: TRansForm
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIC-130-21
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Obesity, Childhood; Obesity, Adolescent
Keywords: Obesity; Time restricted feeding
MeSH Terms: conditions — Pediatric Obesity; Obesity; Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active control (Active Comparator): Participants in this arm will receive the usual treatment for obesity at our hospital, based on lifestyle changes (encouraging a healthy diet and physical activity) for 2 months
  Interventions: Behavioral: Lifestyle intervention
- Time-Restricted Feeding (Experimental): Participants in this arm will receive the usual treatment for obesity at our hospital, based on lifestyle changes (encouraging a healthy diet and physical activity) for 2 months. During this time, participants will have their feeding time restricted to 8 hours per day.
  Interventions: Behavioral: Lifestyle intervention; Behavioral: TRF intervention

INTERVENTIONS:
Behavioral: Lifestyle intervention — Lifestyle intervention (usual treatment for patients with obesity). The behavioral intervention will last for 2 months.
Behavioral: TRF intervention — Food intake restricted to 8 hours per day during the window between 10h and 22h. Time restricted feeding will take place 6 days per week, with the seventh day unrestricted. The intervention will last for 2 months.
  Arms: Time-Restricted Feeding

SUMMARY:
This study will evaluate the effectiveness of a 2-month time-restricted feeding (TRF) intervention in children and adolescents with obesity. The investigators will determine whether the potential beneficial effects of the intervention in this population are maintained over time. Furthermore, potential mechanisms mediating TRF effects will be explored, specifically focusing on the potential role of the gut microbiome and the circadian rhythm.

ELIGIBILITY:
Inclusion Criteria:

* Obesity (BMI z score > 2)

Exclusion Criteria:

* Bariatric surgery
* Spontaneous time-restricted feeding for > 12 hours
* Diabetes with insulin treatment
* Pregnancy
* Intellectual disability
* Under drug treatment with a prescription change in the last 3 months

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 67 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in BMI z score | Baseline, 2 months
  Weight and height will be combined to calculate BMI. The World Health Organization growth charts will be used to calculate BMI z scores.

SECONDARY OUTCOMES:
Change in BMI z score (follow-up) | 1 year, 2 year
  Weight and height will be combined to calculate BMI. The World Health Organization growth charts will be used to calculate BMI z scores.
Change in Adiposity | Baseline, 2 months, 1 year, 2 year
  Adiposity will be measured by bioimpedance
Change in glucose metabolism | Baseline, 2 months, 1 year, 2 year
  Fasting blood test will performed at each time point to analyze glucose metabolism, including glucose, HbA1c, and insulin levels.
Change in lipid profile | Baseline, 2 months, 1 year, 2 year
  Fasting blood test will performed at each time point to analyze the lipid profile, including triglycerides, total cholesterol, LDL-cholesterol, and HDL-cholesterol.
Change in blood pressure | Baseline, 2 months, 1 year, 2 year
  Both systolic and diastolic blood pressure will be measure at every time point
Change in dietary composition | Baseline, 2 months, 1 year, 2 year
  A 4-day food registry will be analyzed at every time point to determine daily energy, macronutrient and micronutrient intake.

OTHER OUTCOMES:
Change in gut microbiota | Baseline, 2 months, 1 year, 2 year
  Fecal samples will be obtained at every time-point and gut microbiota composition analyzed.
Change in circadian rhythm | Baseline, 2 months, 1 year, 2 year
  The circadian rhythm will be measured with an ActTrust actigraph (Condor Instruments) that participants will wear for 2 weeks before each time point.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sant Joan de Deu, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Molina-Giraldo P, Murillo S, Meis L, Sans O, Amat-Bou M, Llobet M, Jimenez-Chillaron JC, Ramon-Krauel M, Lerin C. A time-restricted feeding intervention in children and adolescents with obesity: The TRansForm study protocol. Front Nutr. 2022 Oct 26;9:1026694. doi: 10.3389/fnut.2022.1026694. eCollection 2022. PMID 36386926